CLINICAL TRIAL: NCT02154412
Title: Mechanisms of Arterial Hypotension in Chronic Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Alexander V Ovechkin, MD, PhD, Associate Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 11.0286 Ovechkin
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injury
Keywords: Respiration; Motor control; Blood Pressure; Orthostatic Hypotension
MeSH Terms: conditions — Spinal Cord Injuries; Respiratory Aspiration; Hypotension, Orthostatic | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Respiratory training (Experimental): Subjects will be seated in own wheelchair with head-up tilt. Assembled together, a threshold Positive Expiratory Pressure Device (Respironics, Inc.) & an Inspiratory Muscle Trainer (IMT, Respironics Inc.) with mouthpiece will be used. Subjects will perform maximal inspiratory and expiratory efforts against a pressure load. Participants will be asked to train 45 minutes per day, 5 days per week, for 4 weeks. The training will be initiated with a load equal to 20% of their individual PImax and PEmax with progressive increases as tolerated up to 40% of their baseline PImax or PEmax.
  Interventions: Other: Respiratory Training
- No respiratory training (No Intervention): Participants will not participate in the respiratory muscle training.

INTERVENTIONS:
Other: Respiratory Training — Assembled together using a T-shaped connector, a threshold Positive Expiratory Pressure Device (Respironics, Inc.) & an Inspiratory Muscle Trainer (IMT, Respironics Inc.) with mouthpiece will be used. During inhalation, the subjects will initiate each breath from residual volume (RV) and to sustain the effort until their lungs feel full. During exhalation, the subjects will breathe from total lung capacity and sustain their effort until their lungs feel empty. Participants will be asked to train 45 minutes per day, 5 days per week, for 4 weeks. The training will be initiated with a load equal to 20% of their individual PImax and PEmax with progressive increases as tolerated up to 40% of their baseline PImax or PEmax.
  Arms: Respiratory training

SUMMARY:
This clinical study is designed to investigate the mechanisms of blood pressure regulation and respiratory motor function affected by spinal cord injury (SCI). We hypothesize that impaired blood pressure regulation in individuals with chronic SCI can be improved by restoring respiratory motor function by using Respiratory Motor Training (RMT).

DETAILED DESCRIPTION:
Methods & Procedures

Screening spirometry will be performed with patient sitting in his/her personal wheelchair using BreezeSuite System. Forced Vital Capacity (FVC) & Forced Expiratory Volume in 1 second (FEV1) will be obtained & expressed as the percent of the predicted value for each subject based on a database of neurologically intact individuals with no known pulmonary complaints that was derived based on gender, age, & height. Three acceptable spirograms will be obtained & the result of their best attempt will be used.

Screening Orthostatic Stress Test will be conducted in patient placed on the cardiac chair (Chair Hydraulics). The left hand will be placed in an arm sling & kept at the level of the heart throughout the study. Continuous beat-to beat arterial blood pressure will be acquired from a finger cuff placed around the left middle or index finger (Portapres-2) in supine position & when the participants is moved into the upright seated position. Supine positions will be maintained for 15 min. & upright position will be maintained for 5 min. Baseline values in supine position will be recorded during the last 5-min period just before changing to the upright position. This test will be aborted if subjects become lightheaded or symptomatic of syncope.

Spirometry & Respiratory Muscle Strength Tests: Standard spirometry will be performed in sitting position by using BreezeSuite System (MedGraphics). FVC & FEV1 will be obtained. MP45-36-871-350 Differential Pressure Transducer with UPC 2100 PC card & software (Validyne Engineering) will be used to measure the maximum inspiratory pressure (PImax) & the maximum expiratory pressure (PEmax) in sitting position. The PImax will be measured during maximal inspiratory effort beginning at near residual volume & PEmax will be measured during maximal expiratory effort starting from near total lung capacity. Subjects will be asked to use a three-way valve system with rubber tube as mouthpiece. The pressure meter incorporates a 1.5 mm diameter leak to prevent glottic closure & to reduce buccal muscle contribution during measurements. The assessment will require a sharp, forceful effort be maintained for a minimum of 2 seconds. The maximum pressure will be taken as the highest value that sustained for one second. The maximum value from three maneuvers that varied by less than 20% will be averaged. Participants will be given specific instructions prior to the test & will be verbally coached throughout the spirometry & respiratory muscle strength maneuvers.

Orthostatic Stress Test:

Each participant will be tested in the morning in a quiet, temperature-controlled (~22o C) cardiovascular laboratory. Their diet will be restricted to exclude caffeine, alcohol & foods that are high in fat on the evening prior to & the morning of the study. Participants will be asked to empty their bladder before beginning the study. Continuous arterial BP will be acquired from a finger cuff placed around the left middle or index finger or thumb (Portapres-2;). The left hand will be placed in an arm sling & kept at the level of the heart throughout the study. Manual arterial BP measurements will be taken at the beginning of the supine control period & at the end of the recovery period with a digital blood pressure measurement device. A 3-lead ECG will be placed for ECG monitoring. Rib cage & abdomen kinematics (respiratory kinematics) will be acquired using an inductive plethysmograph. Baseline recording for 15 min. will begin after a 5-minute rest period that will follow subject preparation. At the end of 15-minute recording in the supine position, participants will be passively moved into the upright seated position. This position will be maintained for 15 min. This test will be aborted if subjects become lightheaded or symptomatic of syncope. Hemodynamic variables will be acquired at 1000 Hz using ML880 PowerLab System. ECG, SBP & DBP will be computed from continuous recording, & all variables will be then down-sampled to 5Hz. Beat-to-beat SBP, DBP, RR-interval & HR will be also calculated from acquired continuous BP & ECG. All analyses will be done using Matlab. The Blood flow in the heart will be measured by Cardiac Ultrasound using standard equipment by placing a sensor above the heart.

Blood Catecholamines:

A butterfly catheter will be inserted into an antecubital vein during instrumentation to allow the collection of blood without additional stress to the participant. Eight milliliters of venous blood will be drawn from an antecubital vein at the end of 15-minute supine to assess baseline epinephrine & norepinephrine levels. Blood draw will be repeated at 3 & at the end of 15 min. of upright position to assess quick & steady-state catecholamines responses to orthostatic stress.

Baroreflex evaluation: The last 5 min. of data acquired from each position will be used for further analysis. The beat-to-beat time series of SBP & RR intervals will be scanned for three or more consecutive beats that independently contain increasing & decreasing pressure (SBP+, SBP-) & RR interval (RR+, RR-) with minimum 1 mmHg SBP, & 4 ms RR interval thresholds. If an identified SBP sequence is followed by an identified RR sequence with delay of zero, one, or two beats, those SBP & RR sequences will be assigned as coupled. Only coupled sequences with regression coefficient r>0.90 will be accepted as a baroreflex sequences (BRsq). The mean slope of all BRsq will be calculated & taken as an estimation of baroreflex sensitivity (BRS, ms/mmHg). The numbers of beats involved in SBP ramps & BRsq will be determined at each tilt position. The baroreflex effectiveness index (BEI) will be calculated as the ratio between the total number of BRsq & the total number of SBP ramps.

sEMG protocol: Electrical impulses originate in regulatory neurons, carried via motor nerves, transmit through neuromuscular junction & propagate throughout muscle membranes can be recorded by surface electromyography (sEMG).This physiological test is often relied upon during clinical pulmonary function testing & in research, has been shown to be an accurate reflection of the contractile strength of the respiratory muscles.We will use a multi-muscle sEMG-based measure of motor output from the central nervous system recorded during voluntary motor tasks attempted in the supine position under strictly controlled conditions that was based on Brain Motor Control Assessment (BMCA) principles. The protocol consists of the following voluntary maneuvers followed by 5 min. of quiet breathing: deep breath, PImax task & PEmax task. Each maneuver will be cued by an audible tone & repeated three times. PImax & PEmax during these tasks will be maintained for a minimum of 5 seconds. Airway pressure will be recorded simultaneously with sEMG using a three-way valve system with a pressure transducer as described above. Surface EMG recordings will be accomplished with pairs of recessed, FE9 silver-silver chloride cap surface electrodes (Grass Instruments, W Warwick, RI) centered over the muscle & placed 3 cm apart for each muscle recorded. Skin will be prepared to reduce intra-electrode impedance. Right & left upper portion of pectoralis (PEC), 6th intercostals (IC6), rectus abdominus (RA), & obliquus abdominus (OBL) muscles will be recorded. The ground electrode will be placed over the acromion process. sEMG will be recorded using an Eclipse Neurological Workstation (Axon Systems Inc.). The incoming sEMG signals will be amplified with a gain of 500, filtered at 30-1000 Hz & sampled at 2000 Hz.

Ultrasonic cardiac echography: Standard left ventricular echocardiograms in supine resting state will be obtained measuring end-diastolic diameter (Dd) & the end-systolic diameter (Ds). Ten consecutive beats will be analyzed & the mean will be used for cardiac output (Q) calculations: Q= (Dd)3- (DS)3x HR 35.

Respiratory Muscle Training:

During the training session, subjects will be seated in their personal wheelchair with an approximately 45° head-up tilt. A threshold Positive Expiratory Pressure Device & a threshold Inspiratory Muscle Trainer with flanged mouthpiece will be used for a range of 20 to 41 cm H2O. These devices will be assembled together using a T-shaped connector (Airlife 001504). The participants will be instructed to perform maximal inspiratory & expiratory efforts against a pressure load. During inhalation, the subjects will be instructed to initiate each breath from residual volume (RV) & to sustain the effort until their lungs feel full. During exhalation, the subjects will be instructed to breathe from total lung capacity & sustain their effort until their lungs feel empty. Participants will be asked to train 45 min. per day, 5 days per week, for 4 weeks. The training will be initiated with a load equal to 20% of their individual PImax & PEmax with progressive increases as tolerated up to 40% of their baseline PImax or PEmax. The goal will be to have all patients training at 40% of PImax & PEmax during the last week of the training. An interval training protocol will be used with patients performing six work sets, 5 min. in duration, separated by rest intervals lasting 1-3 min.. A research team member will monitor all training sessions.

Preliminary results showed that RMT will increase FVC, FEV1, PImax & PEmax in experimental subjects compared to pre-training values. The biggest effect is expected for expiratory values (FEV1, & PEmax). One reason for this might be the fact that expiratory function, the most limited after SCI, has bigger window for change. Our results showed that average increase of 8-9% with a sample size of 24-26 patients could reveal a significant difference with a power of 80-86% in all spirometrical values.

Aim 2. Improvement in the BP & mechanisms associated with blood pressure changes were assessed using the low-frequency component of power spectral density of systolic (SBP) & diastolic (DBP) blood pressure values & amount of catecholamines measured in blood levels. Based on preliminary findings small changes are expected in the resting BP values after training. However, after training, the increase in SBP when position is changed to sit-up is expected to be strong with low variability. The calculations showed that even with n=20, the power will be 84% & when n=24, it will be increased to 94%. Changes in DBP are expected to be lower with power of 80% for n=24. Similar values were obtained when low frequency modulations of SBP & DBP were analyzed.

According to this analysis, number of subjects from 20 to 24 will result in significant increase with 87% power. The effectiveness & sensitivity of the baroreflex both improved after training in the preliminary study. After training, in response to the orthostatic stress, a substantial increase in baroreflex responsiveness was obtained & a power of 83% will result with a sample size of 24. The baroreflex sensitivity exhibited much higher variability. If variability remains high in the proposed study, the power of achieving a significant difference from pre-to post-training is 83% with a sample size of 28 patients.

However, a decrease in variability is very likely with a larger sample size & the power increases to 86% with a sample of 24 patients with a 32% decrease in variability.

Based on the results of test-re-test recordings in 10 SCI subjects, the matched number of untrained subjects (n=12) will be enough to form a control group. The deviations from the means were found to be so low, that it would be impossible to reach significance with a reasonable sample size for this group.

ELIGIBILITY:
Inclusion Criteria:

* Non-progressive chronic Spinal Cord Injury (SCI)
* At least 18 years old
* Stable medical condition
* No diseases or conditions that would contraindicate the respiratory muscle training (RMT)
* Not ventilator-dependent for respiration
* At least 15%-deficit in pulmonary function outcome measures
* Orthostatic hypotension

Exclusion Criteria:

* Major cardiovascular or pulmonary disease
* Endocrine disorders
* Malignancy
* Pregnancy (no pregnancy test or birth control regimen will be required)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Pulmonary function test | Before and after 20 sessions of RMT
  Standard spirometry measures in percent predicted values

SECONDARY OUTCOMES:
Blood pressure change measurement | Before and after 20 sessions of RMT
  Beat-to-beat blood pressure in mmHg
Maximum airway pressure | Before and after 20 sessions of RMT
  Airway pressure in cm H2O

OTHER OUTCOMES:
Cardiac ultrasound | Before and After 20 RMT sessions
  Blood flow in the heart will be measured by licensed clinical personnel using standard equipment by placing a sensor above the heart.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Ovechkin, PhD, Principal Investigator — University of Louisville
Locations (1):
- Frazier Rehabilitation and Neuroscience Institute, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeVivo MJ, Krause JS, Lammertse DP. Recent trends in mortality and causes of death among persons with spinal cord injury. Arch Phys Med Rehabil. 1999 Nov;80(11):1411-9. doi: 10.1016/s0003-9993(99)90252-6. PMID 10569435
- [Background] Krassioukov A. Autonomic function following cervical spinal cord injury. Respir Physiol Neurobiol. 2009 Nov 30;169(2):157-64. doi: 10.1016/j.resp.2009.08.003. Epub 2009 Aug 12. PMID 19682607
- [Background] Teasell RW, Arnold JM, Krassioukov A, Delaney GA. Cardiovascular consequences of loss of supraspinal control of the sympathetic nervous system after spinal cord injury. Arch Phys Med Rehabil. 2000 Apr;81(4):506-16. doi: 10.1053/mr.2000.3848. PMID 10768544
- [Background] Claydon VE, Krassioukov AV. Orthostatic hypotension and autonomic pathways after spinal cord injury. J Neurotrauma. 2006 Dec;23(12):1713-25. doi: 10.1089/neu.2006.23.1713. PMID 17184183
- [Background] Bernard PL, Mercier J, Varray A, Prefaut C. Influence of lesion level on the cardioventilatory adaptations in paraplegic wheelchair athletes during muscular exercise. Spinal Cord. 2000 Jan;38(1):16-25. doi: 10.1038/sj.sc.3100956. PMID 10762193
- [Background] Frankel HL, Coll JR, Charlifue SW, Whiteneck GG, Gardner BP, Jamous MA, Krishnan KR, Nuseibeh I, Savic G, Sett P. Long-term survival in spinal cord injury: a fifty year investigation. Spinal Cord. 1998 Apr;36(4):266-74. doi: 10.1038/sj.sc.3100638. PMID 9589527
- [Background] Garshick E, Kelley A, Cohen SA, Garrison A, Tun CG, Gagnon D, Brown R. A prospective assessment of mortality in chronic spinal cord injury. Spinal Cord. 2005 Jul;43(7):408-16. doi: 10.1038/sj.sc.3101729. PMID 15711609
- [Background] De Troyer A, Estenne M, Heilporn A. Mechanism of active expiration in tetraplegic subjects. N Engl J Med. 1986 Mar 20;314(12):740-4. doi: 10.1056/NEJM198603203141203. PMID 3951503
- [Background] Winslow C, Rozovsky J. Effect of spinal cord injury on the respiratory system. Am J Phys Med Rehabil. 2003 Oct;82(10):803-14. doi: 10.1097/01.PHM.0000078184.08835.01. PMID 14508412
- [Background] Laffont I, Durand MC, Rech C, De La Sotta AP, Hart N, Dizien O, Lofaso F. Breathlessness associated with abdominal spastic contraction in a patient with C4 tetraplegia: a case report. Arch Phys Med Rehabil. 2003 Jun;84(6):906-8. doi: 10.1016/s0003-9993(02)04898-0. PMID 12808547
- [Background] Walter JS, Sacks J, Othman R, Rankin AZ, Nemchausky B, Chintam R, Wheeler JS. A database of self-reported secondary medical problems among VA spinal cord injury patients: its role in clinical care and management. J Rehabil Res Dev. 2002 Jan-Feb;39(1):53-61. PMID 11926327
- [Background] Claydon VE, Steeves JD, Krassioukov A. Orthostatic hypotension following spinal cord injury: understanding clinical pathophysiology. Spinal Cord. 2006 Jun;44(6):341-51. doi: 10.1038/sj.sc.3101855. Epub 2005 Nov 22. PMID 16304564